CLINICAL TRIAL: NCT04961658
Title: Advanced Mesenchymal Enhanced Cell THerapY for SepTic Patients
Acronym: AMETHYST
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding Decision
Sponsor: Northern Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT-GEM-001
Record Dates: First submitted 2021-06-24; First posted 2021-07-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Septic Shock
Keywords: Sepsis; Bacteria; Septic Shock; Mesenchymal Stromal Cells; Inflammation; Mesenchymal Stem Cells; Infection
MeSH Terms: conditions — Shock, Septic; Sepsis; Inflammation; Infections

STUDY DESIGN:
Intervention Model Description: A dose-escalation study evaluating GEM00220 cell therapy in 4 cohorts with 3 subjects per cohort. Study will proceed from lower dose to next higher dose if no safety concerns are observed in each cohort. If no safety issues are identified, we will continue to the Phase 1b trial.
  Phase 1b: A single-arm, open-label extension of the Phase 1a trial to assess early signs of efficacy (major morbidity and mortality). The Phase 1b trial will enroll up to 9 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Arm - Dose Cohort 1 (Experimental): Participants will receive a single dose of GEM00220 at 15 million cells
  Interventions: Biological: GEM00220
- Treatment arm - Dose Cohort 2 (Experimental): Participants will receive a single dose of GEM00220 at 60 million cells
  Interventions: Biological: GEM00220
- Treatment arm - Dose Cohort 3 (Experimental): Participants will receive a single dose of GEM00220 at 150 million cells
  Interventions: Biological: GEM00220
- Treatment arm - Dose Cohort 4 (Experimental): Participants will receive two doses of GEM00220 at 150 million cells each, seperated by 24 hours
  Interventions: Biological: GEM00220

INTERVENTIONS:
Biological: GEM00220 — Cryopreserved allogeneic, enhanced MSCs administered as a single intravenous infusion

SUMMARY:
Bacterial sepsis occurs in patients with severe infections. The condition is caused by toxic substances (toxins) released from bacteria and the patient's elevated inflammatory response to those toxins. In preclinical studies, human mesenchymal stromal cells (MSCs) have been proven to modulate host inflammation in infections, including sepsis. The purpose of the Phase I, open label, dose escalation safety trial is to determine whether escalating doses of enhanced MSCs (GEM00220) are safe and well tolerated in patients with septic shock.

DETAILED DESCRIPTION:
This trial consists of 2 sequential parts using the same trial infrastructure:

Phase 1a: A dose escalating and safety trial with pre-defined stopping rules for safety. Up to 12 participants will receive a single infusion of GEM00220. If no safety issues are identified, we will continue to the Phase 1b trial at the maximum feasible tolerated dose.

Phase 1b: A single-arm, open-label extension of the Phase 1a trial to assess early signs of efficacy (major morbidity and mortality). The Phase 1b trial will enroll up to 9 participants to assess early signals of benefit on mortality and major morbidity in a high risk, high mortality population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients age 18 years and older
2. Receipt of appropriate antibiotics for the suspected/confirmed bacterial sepsis as the main diagnosis according to the opinion of the treating staff physician.
3. Hypotension documented within 48 hours prior to enrolment that requires the institution and ongoing use of vasopressor agents (phenylephrine, norepinephrine, vasopressin, epinephrine, or dopamine >5 mcg/kg/min) for at least 3 hours within 24 hours prior to infusion, despite adequate fluid resuscitation in the opinion of the qualified investigator.
4. At least 1 other new organ dysfunction defined by the following:

   1. Renal: Acute kidney injury with creatinine ≥ 150 µmol/L, or ≥ 1.5x the upper limit of normal or the known baseline creatinine, or < 0.5 ml/kg/hr urine output for 6 hours despite adequate fluid resuscitation or requirement for new renal replacement therapy (patients on chronic hemodialysis or peritoneal dialysis must meet one of the other organ dysfunction criteria)
   2. Respiratory: Need for invasive mechanical ventilation or a P/F ratio < 250
   3. Hematological: Platelets < 100 x10^9/L, or a drop of 50 x10^9/L in the 3 days prior to enrollment
   4. Metabolic Acidosis: Arterial pH < 7.30 in association with base deficit > 5 mmol/L OR a lactate >/= to 3.0 mmol/L

Exclusion Criteria:

1. Pregnant or lactating
2. Currently receiving extracorporeal life support
3. Major surgery within this hospitalization and not prophylactically anticoagulated
4. Documented history of a hypercoagulable state (eg Factor V Leiden) or heparin-induced thrombocytopenia (HIT)
5. Body Mass Index (BMI) > 35
6. Documented COVID-19 (SARS-CoV2) within 30 days
7. Documentation of viral lung infection as the primary diagnosis (e.g. influenza infection, respiratory syncytial virus (RSV) infection, or other laboratory-confirmed viral lung infection)
8. Presence of any active malignancy (other than non-melanoma skin cancer) that required treatment within the past year
9. Documented history of severe heart failure with a New York Heart Association Functional Class of III or IV, or severe ischemic heart disease with a Canadian Cardiovascular Society angina class score of III or IV
10. Documented history of moderate to severe chronic liver disease (Childs-Pugh Score > 12)
11. Documented history of peripheral vascular disease with a Rutherford classification greater than Grade I, Category 2: moderate claudication
12. Severe chronic respiratory disease with a baseline PaCO2 > 50 mm Hg or the use of home oxygen
13. Documented deep venous thrombosis or pulmonary embolism
14. Chronic immunosuppression (any chronic immunotherapy including daily oral steroid use >6months)
15. Documented, uncontrolled HIV infection or end stage HIV/AIDS with CD4+ T-cell counts <50 cells/mm^3, history of hepatitis B, untreated hepatitis C, or active tuberculosis
16. Concurrent use of immunomodulatory biologic drugs or TNF-α inhibitors
17. Participation in another interventional study involving an investigational new drug within 30 days prior to enrolment
18. Moribund patient not expected to survive 24 hours
19. Patient, surrogate, or physician not committed to full support (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
The safety of GEM00220 will be assessed by monitoring adverse events | Baseline to 28 days
Maximum Feasible Tolerated Dose | Baseline to 28 days
  The highest dose which does not meet any of the pre-defined stopping criteria

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Markham Stouffville Hospital - Oak Valley Health, Markham, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No